CLINICAL TRIAL: NCT01541111
Title: Evaluation of Analgesic Effect of Magnesiun Associated With Morphine for Cancer Pain Relief
Brief Title: Magnesium Associated With Morphine for Cancer Pain Relief
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Federal University of São Paulo (Other)
Responsible Party: Principal Investigator, Rioko Kimiko Sakata, PhD, Federal University of São Paulo
Allocation: Not Applicable | Model: Single Group | Masking: Double | Purpose: Treatment
Other Study IDs: CEP0153/09
Record Dates: First submitted 2012-02-17; First posted 2012-02-29 (Estimated); Last update posted 2015-07-28 (Estimated); Status verified 2015-07

CONDITIONS: Cancer-related Problem/Condition
Keywords: Cancer pain; Magnesiun
MeSH Terms: conditions — Cancer Pain | interventions — GluN2C-2D antagonist UBP145

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (1):
- Magnesiun, pain relief, sugar pills (Other): Magnesiun 75mg po each 12h pain relief Sugar pills po each 12h
  Interventions: Drug: Magnesiun

INTERVENTIONS:
Drug: Magnesiun — 75mg pills; each 12h; 12wk
  Other Names: NMDA receptor antagonist

SUMMARY:
This study is an evaluation of the analgesic effect of magnesium associated with morphine in patients with cancer pain.

DETAILED DESCRIPTION:
The study is prospective, randomized, double-blind. The patients will be allocated into two groups. After approval by the Ethics Committee and signed informed consent, 40 patients, aged > 18 years of both genders with cancer pain, will be studied.

The patients in group 1 (n = 20) will receive a dose of magnesium sulfate (65 mg) po twice daily. Patients in Group 2 (n = 20) will receive placebo twice a day. The Mg and placebo capsules are identical. Everyone will receive morphine as needed.

Will be recorded: tumor location, factors which worsen the pain, quality of pain. Pain intensity will be assessed by numerical scale from zero to 10 at T0 (first visit) and after 1, 2, 3. and 4wk.

The patient will note the intensity of pain and side effects at home. Functional performance assessment will bes done by the Karnofsky Performance Status Scale. Quality of life will be assessed by the QLQ-c30.

ELIGIBILITY:
Inclusion Criteria:

* After approval by the Ethics Committee and signed informed consent,
* 40 patients, > 18 years, with cancer pain, and taking morphine (third step of the analgesic ladder recommended by WHO) were studied

Exclusion Criteria:

* Were excluded from the study patients with hypersensitivity to drugs and pregnant

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Actual)
Dates: Start 2011-01; Primary Completion 2014-03 (Actual); Study Completion 2014-03 (Actual)

PRIMARY OUTCOMES:
Pain relief | 12 wk

SECONDARY OUTCOMES:
Morphine dose | 12 wk

CONTACTS AND LOCATIONS:
Overall Officials: Rioko K Sakata, MD, PhD, Study Director — Universidade Federal de São Paulo
Locations (1):
- Universidade Federal de São Paulo, São Paulo, São Paulo, Brazil